CLINICAL TRIAL: NCT02564861
Title: A Phase I, Double-Blind, Randomised, Placebo Controlled, Multiple-Dose Study to Assess Safety, Tolerability and Pharmacokinetics of DS-1971a in Healthy Male and Female Subjects
Brief Title: Multiple Dose Study of D1971a in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: DS1971-A-E106; 2015-002885-22 (EudraCT Number)
Record Dates: First submitted 2015-09-28; First posted 2015-10-01 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Healthy
Keywords: pharmacokinetics
MeSH Terms: interventions — DS-1971a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- DS-1971a (Low Dose) (Experimental): Participants in Cohort 1 who receive a low dose of DS 1971a in an oral suspension
  Interventions: Drug: DS-1971a
- DS-1971a (Mid dose) (Experimental): Participants in Cohort 2 who receive a mid dose of DS 1971a in an oral suspension
  Interventions: Drug: DS-1971a
- DS-1971a (High dose) (Experimental): Participants in Cohort 3 who receive a high dose of DS 1971a in an oral suspension
  Interventions: Drug: DS-1971a
- Pooled placebo (Experimental): Participants in Cohort 1, 2 or 3 who receive matching DS-1971a Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DS-1971a — DS 1971a is supplied as a powder or crystals and will be given as an oral suspension
  Arms: DS-1971a (High dose); DS-1971a (Low Dose); DS-1971a (Mid dose)
Drug: Placebo — Placebo matching DS-1971a suspension
  Arms: Pooled placebo

SUMMARY:
This is a randomised, double-blind, placebo-controlled multiple dose study designed to explore the safety, tolerability and PK of DS-1971a following oral administration over 14 days to healthy male and female subjects. Each participant receives lidocaine as a local anaesthetic before inserting the intravenous cannula.

DETAILED DESCRIPTION:
Within strictly defined limits, the protocol permits the dose escalation committee to amend the dose escalation rules, doses proposed in the study protocol and to change the timing of or to add additional assessments following review of the safety, tolerability and plasma DS-1971a concentration data. The decisions to change the doses will be documented in the minutes of the dose escalation committee.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects aged 18 years to 65 years.
* A body mass index (BMI) in the range 18 kg/m2 to 30 kg/m2, inclusive, and weighing between 50 kg and 100 kg, inclusive at screening. BMI is calculated as weight [kg]/(height [m])2.
* Female subjects must be of non-childbearing potential as follows:

  * Must be postmenopausal (the last menstrual period was at least 12 months before Screening, and a follicle stimulating hormone [FSH] test at Screening confirms postmenopausal status); or
  * Must be surgically sterile having undergone hysterectomy, bilateral oophorectomy, bilateral salpingectomy and/or bilateral tubal ligation.
* Willing to comply with all study restrictions, including the use of contraception, concomitant medication, and dietary and lifestyle restrictions.
* Sufficient intelligence to understand the nature of the study and any hazards of participating in it. Ability to communicate satisfactorily with the Investigator and to participate in, and comply with requirements of, the entire study.
* Have given written consent to participate in the study after reading the ICF, and after having the opportunity to discuss the study with the Investigator or his delegate.
* Have given written consent to have his/her data entered into The Over volunteering Prevention System.

Exclusion Criteria:

* Clinically relevant abnormal history, physical findings, ECG findings, or laboratory values that could interfere with the objectives of the study or compromise the safety of the subject.
* Presence or history of acute or chronic illness, including (but not limited to) liver or kidney disease, hypertension, seizures, or any known impairment of endocrine, or other specific body-organ dysfunction.
* History of serious reaction to any medicine.
* Presence or history of malignant disease.
* Acute or chronic infectious disease, including human immunodeficiency virus (HIV), hepatitis B virus (HBV) or C virus (HCV) infection.
* Surgery (eg, stomach bypass) or medical condition that might affect how the body handles or absorbs medicines.
* Significant illness within 4 weeks before the first dose of study medication.
* Participation in another clinical study of a new chemical entity or a prescription medicine within the previous 3 months, or unwilling to abstain from participating in other clinical trials during the study and for 3 months after receipt of study medication.
* Blood pressure (BP) and heart rate in semi-supine position at the Screening examination outside the ranges 90 mmHg to 140 mmHg systolic, 40 mmHg to 90 mmHg diastolic; heart rate < 40 beats/min to > 100 beats/min. Subjects with Stage 1 hypertension (systolic 140 mmHg to 160 mmHg; diastolic 90 mmHg to 100 mmHg) may be enrolled provided they do not have evidence of end-organ damage, diabetes or a 10 year cardiovascular risk > 20%.
* Abnormal ECG waveform morphology at Screening that would preclude accurate measurement of the uncorrected QT interval (QT) duration.
* QT interval for heart rate corrected using QTcF interval duration > 430 ms for men or > 450 ms for women, obtained as an average from the measurements on duplicate Screening ECGs over a brief recording period.
* Estimated glomerular filtration rate (eGFR) < 80 mL/min/1.73m2 (based on Modification of Diet in Renal Disease [MDRD] equation) or an absolute creatinine value outside the normal range.
* Use of any prescription or over the counter (OTC) medications, or herbal remedies (such as St John's wort), known to be strong inhibitors or strong inducers of cytochrome (CYP) enzymes (also known as CYP P450 enzymes) during the 30 days before the first dose of study medication; use of any other prescription or OTC medicine (with the exception of acetaminophen (paracetamol)), including dietary supplements or herbal remedies, during the 7 days before the dose of study medication.
* Pregnant or breastfeeding women.
* Consumption of certain foods or beverages before the first dose and throughout the study period.
* Loss of more than 400 mL blood or donation of blood, plasma, platelets, or any other blood components during the 3 months before the first dose of study medication, or unwilling to abstain from doing so during the study and for 3 months after receipt of study medication.
* Abuse of drugs or alcohol during the 2 years before the first dose of study medication, or intake of more than 21 units of alcohol weekly for male subjects and 14 units of alcohol weekly for female subjects.
* Use of tobacco products or nicotine-containing products during the 3 months before the first dose of study medication and during the study.
* Evidence of drug or alcohol abuse at screening or admission.
* Likely possibility that the volunteer will not cooperate with the requirements of the protocol.
* Objection by General Practitioner (GP) to the volunteer entering the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with at least one Treatment Emergent Adverse Event (TEAEs) | 14 days
  TEAEs are adverse events that began or got worse after treatment began. Clinically significant changes in laboratory tests and/or physical examinations are considered adverse events.

SECONDARY OUTCOMES:
Cmax of DS-1971a | Day 1 and Day 14
  Cmax is the highest concentration of the drug in the blood
Tmax of DS-1971a | Day 1 and Day 14
  Tmax is the time it takes for Cmax to be reached
Area Under Curve at steady state (AUCtau) of DS-1971a | Day 1 and Day 14
  AUCtau is the area under the plasma concentration-time curve at steady state. In pharmacokinetics, steady state refers to the situation where the overall intake of a drug is about even with the rate it is being eliminated from the body.
Area under the Curve (additional measures) for DS-1971a | Day 1 and Day 14
  Additional AUC measures include AUC0-24 (to 24 hours), AUClast (to the last observable measure), AUC0-inf (to infinity), and AUCextr (from AUClast to infinity)
Tmax of DS-1971a metabolites M1 and M2 | Day 1 and Day 14
  Tmax of metabolites M1 and M2 characterized by Tmax
Cmax of DS-1971a metabolites M1 and M2 | Day 1 and Day 14
  Cmax of metabolites M1 and M2 characterized by Cmax
AUC of DS-1971a metabolites M1 and M2 | Day 1 and Day 14
  AUC measures include AUCtau, AUC0-24, AUClast, AUC0-inf

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (1):
- Mammersmith Medicines Research Ltd., London, United Kingdom